CLINICAL TRIAL: NCT05974683
Title: A Study of Two Different Treatment Strategies in IgG4-related Disease Patients With Re-elevation of Serum IgG4 Level During Maintenance Remission Period: a Randomized Double Blind Placebo Controlled Multicenter Study
Brief Title: Treatment Strategies in IgG4-RD Patients With Re-elevation of Serum IgG4 Level During Maintenance Remission Period
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Beijing Friendship Hospital (Other); Tongji Hospital (Other)
Responsible Party: Principal Investigator, Wen Zhang, Professor, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IgG4 re-elevation treatment
Record Dates: First submitted 2023-07-05; First posted 2023-08-03 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-07

CONDITIONS: Autoimmune Diseases
Keywords: Immunoglobulin G4-Related Disease; Drug therapy; Relapse
MeSH Terms: conditions — Autoimmune Diseases; Immunoglobulin G4-Related Disease; Recurrence | interventions — Mycophenolic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Basic Maintenance Treatment (Placebo Comparator): Continue use of current basic maintenance treatment of IgG4-RD plus placebo, Follow-up intervals: week 4, week 12, week 24, week 36, week 52
  Interventions: Drug: placebo
- Enhancement Treatment (Active Comparator): Use low dose mycophenolate mofetil (0.5g per day) as an add-on therapy of current basic maintenance treatment of IgG4-RD, Follow-up intervals: week 4, week 12, week 24, week 36, week 52
  Interventions: Drug: mycophenolate mofetil

INTERVENTIONS:
Drug: placebo — Continue use of current basic maintenance treatment of IgG4-RD plus placebo, Follow-up intervals: week 4, week 12, week 24, week 36, week 52
  Arms: Basic Maintenance Treatment
Drug: mycophenolate mofetil — Use low dose mycophenolate mofetil (0.5g per day) as an add-on therapy of current basic maintenance treatment of IgG4-RD, Follow-up intervals: week 4, week 12, week 24, week 36, week 52
  Arms: Enhancement Treatment

SUMMARY:
This study has been designed as a 52-week, randomized double blind placebo controlled multicenter clinical trial. The study aims to compare the efficacy and safety of two treatment strategies in IgG4-RD patients with re-elevation of serum IgG4 level during maintenance remission period: basic maintenance treatment group (continue use of basic maintenance treatment of IgG4-RD) and enhanced treatment group (use low dose mycophenolate mofetil as an add-on therapy of basic maintenance treatment of IgG4-RD).

DETAILED DESCRIPTION:
108 IgG4-RD patients with re-elevation of serum IgG4 level to ≥30% of baseline serum IgG4 level during maintenance remission period are to be enrolled in this study after screening period, and then double blind randomly in an 1:1 ratio into two groups: basic maintenance treatment group (continue use of basic maintenance treatment of IgG4-RD plus placebo) and enhanced treatment group (use low dose mycophenolate mofetil as an add-on therapy of basic maintenance treatment of IgG4-RD). The follow-up period will be 52 weeks. During the follow-up period, clinical evaluations, laboratory tests, image examinations and IgG4-RD responder index (RI) will be recorded. The primary endpoint is the difference of relapse rate between two groups at 52 weeks. Meanwhile, this study will also explore and study different biomarkers in IgG4-RD patients, to better understand the mechanisms, as well as prognostic factors of IgG4-RD.

ELIGIBILITY:
Inclusion Criteria:

* 1. Fulfillment of the 2019 American College of Rheumatology/European League against Rheumatology (ACR/EULAR) IgG4-related disease classification criteria or the 2020 revised comprehensive diagnostic (RCD) criteria for IgG4-RD.
* 2. Age between 18 and 70 years.
* 3. Elevation of baseline serum IgG4 level (>1400mg/L).
* 4. Major organ involvement, including but not limited to autoimmune pancreatitis, retroperitoneal fibrosis, sclerosing cholangitis, IgG4-related Castleman disease, and involvement of the lungs, kidney, nasal sinus, and central nervous system.
* 5. Re-elevation of serum IgG4 level to ≥30% of baseline serum IgG4 level during maintenance remission period, with no evidence of relapse.
* 6. Written informed consent signed.
* 7. Agreed to take highly effective contraceptive procedures from signing of informed consent till 6 months after the end of last visit.

Exclusion Criteria:

* 1. Patients with an IgG4-RD Responder Index ≥ 2 points of any organ system.
* 2. IgG4-RD patients without major organ involvement.
* 3. Patients with severe or active infections, including but not limited to HIV, HCV, HBV, TB.
* 4. Patients with malignancies or a history of malignancies within 5 years, except:

  1. Patients with adenocarcinoma in situ (AIS) of the cervix who have received curative treatment for at least 12 months before screening.
  2. Patients with cutaneous basal or squamous cell carcinoma who have received curative treatment.
  3. Patients with prostate cancer, who have received radical prostatectomy or definitive radiotherapy for over 3 years, with no sign of relapse or ongoing treatment
* 5. Patients with immunodeficiency diseases.
* 6. Patients with severe cardiovascular, respiratory, endocrine, gastrointestinal, hematological, neuropsychological, or constitutional comorbidities; or at risk of unacceptable complications, or having confounding factors in safety and explanation of results according to the evaluations from investigators.
* 7. Patients with other rheumatic diseases, including but not limited to rheumatoid arthritis, systemic lupus erythematosus, systemic vasculitis, sarcoidosis; or other mimickers of IgG4-RD, including but not limited to Rosai-Dorfman disease, Castleman disease.
* 8. Participating in any other clinical trials with drug interventions.
* 9. A history of alcohol or drug abuse, possibly harming patient's safety, compliance, or evaluation of study's safety or other necessary aspects according to the evaluations from investigators.
* 10. Women during pregnancy, lactation, or planning of pregnancy within 6 months of the last visit of the study.
* 11. Meeting any of the following blood test finding on screening:

  1. Hemoglobin level < 7.5g/dL.
  2. neutrophil count < 1.0×10^9/L.
  3. Platelet count < 100×10^9/L.
  4. Alanine aminotransferase (ALT) > 2 × upper limit number (ULN).
  5. Aspartate aminotransferase (AST) > 2 × ULN.
  6. Total Bilirubin (TBil) > 2 × ULN.
  7. Estimated glomerular filtration rate (eGFR) < 30ml/(min·1.73m^2), calculated using the Modification of Diet in Renal Disease (MDRD) study equation by the National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The difference of relapse rate of IgG4-RD between two groups in week 52. | 52 weeks
  The primary endpoint is the difference of relapse rate between two groups at 52 weeks. The definition of relapse: elevation of IgG4-RD Responder Index ≥ 2 points; new organ involvement or recurrence, with or without elevation of serum IgG4 levels.

SECONDARY OUTCOMES:
The difference of relapse rate of IgG4-RD between two groups in the week 12. | 12 weeks
The difference of relapse rate of IgG4-RD between two groups in the week 24 | 24 weeks
The difference of relapse rate of IgG4-RD between two groups in the week 36. | 36 weeks
The time and duration of relapse | 52 weeks
The changes of IgG4-RD Responder Index at week 52 | 52 weeks
The changes of serum IgG level at week 52 | 52 weeks
The changes of serum IgG4 level at week 52 | 52 weeks
The changes of erythrocyte sedimentation rate at week 52 | 52 weeks
The changes of serum C-reactive protein level at week 52 | 52 weeks
Adverse effect events | 52 weeks
The changes of Physician Global Assessment score at week 52 | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Wen Zhang, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Zhang W, Stone JH. Management of IgG4-related disease. Lancet Rheumatol. 2019 Sep;1(1):e55-e65. doi: 10.1016/S2665-9913(19)30017-7. Epub 2019 Aug 28. PMID 38229361
- [Background] Wallace ZS, Naden RP, Chari S, Choi HK, Della-Torre E, Dicaire JF, Hart PA, Inoue D, Kawano M, Khosroshahi A, Lanzillotta M, Okazaki K, Perugino CA, Sharma A, Saeki T, Schleinitz N, Takahashi N, Umehara H, Zen Y, Stone JH; Members of the ACR/EULAR IgG4-RD Classification Criteria Working Group. The 2019 American College of Rheumatology/European League Against Rheumatism classification criteria for IgG4-related disease. Ann Rheum Dis. 2020 Jan;79(1):77-87. doi: 10.1136/annrheumdis-2019-216561. Epub 2019 Dec 3. PMID 31796497
- [Background] Lin W, Lu S, Chen H, Wu Q, Fei Y, Li M, Zhang X, Tian X, Zheng W, Leng X, Xu D, Wang Q, Shen M, Wang L, Li J, Wu D, Zhao L, Wu C, Yang Y, Peng L, Zhou J, Wang Y, Sha Y, Huang X, Jiao Y, Zeng X, Shi Q, Li P, Zhang S, Hu C, Deng C, Li Y, Zhang S, Liu J, Su J, Hou Y, Jiang Y, You X, Zhang H, Yan L, Zhang W, Zhao Y, Zeng X, Zhang F, Lipsky PE. Clinical characteristics of immunoglobulin G4-related disease: a prospective study of 118 Chinese patients. Rheumatology (Oxford). 2015 Nov;54(11):1982-90. doi: 10.1093/rheumatology/kev203. Epub 2015 Jun 22. PMID 26106212
- [Background] Umehara H, Okazaki K, Kawa S, Takahashi H, Goto H, Matsui S, Ishizaka N, Akamizu T, Sato Y, Kawano M; Research Program for Intractable Disease by the Ministry of Health, Labor and Welfare (MHLW) Japan.. The 2020 revised comprehensive diagnostic (RCD) criteria for IgG4-RD. Mod Rheumatol. 2021 May;31(3):529-533. doi: 10.1080/14397595.2020.1859710. Epub 2021 Jan 28. PMID 33274670
- [Background] Khosroshahi A, Wallace ZS, Crowe JL, Akamizu T, Azumi A, Carruthers MN, Chari ST, Della-Torre E, Frulloni L, Goto H, Hart PA, Kamisawa T, Kawa S, Kawano M, Kim MH, Kodama Y, Kubota K, Lerch MM, Lohr M, Masaki Y, Matsui S, Mimori T, Nakamura S, Nakazawa T, Ohara H, Okazaki K, Ryu JH, Saeki T, Schleinitz N, Shimatsu A, Shimosegawa T, Takahashi H, Takahira M, Tanaka A, Topazian M, Umehara H, Webster GJ, Witzig TE, Yamamoto M, Zhang W, Chiba T, Stone JH; Second International Symposium on IgG4-Related Disease. International Consensus Guidance Statement on the Management and Treatment of IgG4-Related Disease. Arthritis Rheumatol. 2015 Jul;67(7):1688-99. doi: 10.1002/art.39132. No abstract available. PMID 25809420
- [Background] Yunyun F, Yu P, Panpan Z, Xia Z, Linyi P, Jiaxin Z, Li Z, Shangzhu Z, Jinjing L, Di W, Yamin L, Xiaowei L, Huadan X, Xuan Z, Xiaofeng Z, Fengchun Z, Yan Z, Wen Z. Efficacy and safety of low dose Mycophenolate mofetil treatment for immunoglobulin G4-related disease: a randomized clinical trial. Rheumatology (Oxford). 2019 Jan 1;58(1):52-60. doi: 10.1093/rheumatology/key227. PMID 30124952
- [Background] Peng Y, Li JQ, Zhang PP, Zhang X, Peng LY, Chen H, Zhou JX, Zhang SZ, Yang HX, Liu JJ, Guo HF, Li J, Zhang X, Zhao Y, Zeng XF, Zhang FC, Fei YY, Zhang W. Clinical outcomes and predictive relapse factors of IgG4-related disease following treatment: a long-term cohort study. J Intern Med. 2019 Nov;286(5):542-552. doi: 10.1111/joim.12942. Epub 2019 Jun 17. PMID 31121062
- [Background] Liu Z, Peng Y, Li J, Lu H, Peng L, Zhou J, Zhou S, Huang C, Wang M, Zhu L, Chen H, Wang L, Fei Y, Zhao Y, Zeng X, Zhang W. Prediction of new organ onset in recurrent immunoglobulin G4-related disease during 10 years of follow-up. J Intern Med. 2022 Jul;292(1):91-102. doi: 10.1111/joim.13477. Epub 2022 Apr 13. PMID 35419810